CLINICAL TRIAL: NCT06374251
Title: Can Narrative Medicine Methods Improve Well-Being in Patients With GI Malignancies
Brief Title: Narrative Medicine for Improving Well-Being in Patients With Gastrointestinal Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0S-23-2; NCI-2023-08890 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-23-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Malignant Digestive System Neoplasm
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (narrative medicine sessions) (Experimental): Patients participate in narrative medicine sessions over 60 minutes Q2W for 3 sessions.
  Interventions: Procedure: Discussion; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Procedure: Discussion — Participate in narrative medicine sessions
  Other Names: Discuss
Other: Interview — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial assesses whether narrative medicine methods may improve the sense of well-being among gastrointestinal (GI) (digestive system) cancer patients. Narrative medicine is a clinical approach where providers can use a patient's own narrative (perspective) of their illness to promote healing and resilience. By applying narrative medicine's main tool, close reading, to clinical practice, clinicians learn to listen and attend to patients more deeply. This allows for freer communication and the creation of a healthcare encounter that centers on the psychological and emotional well being of the patient in addition to their medical conditions. Narrative medicine can include close reading, creative or reflective writing, and discussion. These methods may help patients with GI cancer to reflect on their life stories, both inside and outside of their illness experience, and help them gather skills to optimize their well-being.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of implementing narrative medicine tools in serial workshops with patients with malignancy.

II. To determine if narrative medicine interventions improve markers and expressions of well-being.

DESCRIPTIVE OBJECTIVES:

I. To estimate changes in markers and expressions of well-being after 3 sessions of narrative medicine intervention.

II. To determine, through qualitative methods, if patients find benefit from the intervention regarding their well-being.

III. To decide whether to expand these kinds of interventions to a larger study with control group.

OUTLINE:

Patients participate in narrative medicine sessions over 60 minutes once every 2 weeks (Q2W) for 3 sessions.

After completion of study intervention, patients are followed up at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of gastrointestinal malignancy actively receiving infusional therapy for cancer.
* Age >= 18 years.
* English speaking with ability to participate in reading and writing questionnaires and implementation tools.
* Performance Status =< Eastern Cooperative Oncology Group (ECOG) 3.

Exclusion Criteria:

* Altered mental status or other cognitive impairment, organic or drug induced that would limit ability to participate in the evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete the narrative medicine sessions | Up to 3 months
  To determine the intervention feasibility, the number of participants who complete the narrative medicine sessions will be tracked.
Change in well-being scores | Up to 3 months
  Will be evaluated using the Edmonton Symptom Assessment System-Revised Version (ESAS-r). The total score ranges from 0 to 10, with a higher score indicating worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Eve L Makoff, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States